CLINICAL TRIAL: NCT01493089
Title: A Phase III, Multi-centre, Double-blind, Double-dummy, Randomised, Study to Assess the Superiority of Zegerid® 20 mg vs. Losec® 20 mg in the Rapid Relief of Heartburn Associated With GERD as on Demand Therapy
Brief Title: Phase III Study Comparing Zegerid® With Losec® for the Relief of Heartburn Associated With Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZEG-01/2010 (GERD)
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — omeprazole, sodium bicarbonate drug combination; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zegerid (Experimental): Treatment of heartburn with Zegerid
  Interventions: Drug: Zegerid
- Losec (Active Comparator): Treatment of heartburn with Losec
  Interventions: Drug: Losec

INTERVENTIONS:
Drug: Zegerid — 20 mg Zegerid suspension to be taken when heartburn occurs. Maximum one dose per day on 3 out of 14 days.
  Arms: Zegerid
Drug: Losec — 20 mg Losec capsule to be taken when heartburn occurs. Maximum one dose per day on 3 out of 14 days.
  Arms: Losec

SUMMARY:
Heartburn is the main symptom of Gastroesophageal Reflux Disease (GERD), which, accompanied by acid regurgitation and other symptoms, has a substantial negative impact on a patients' quality of life. Although a number of treatment options are available, a more effective therapy is still required. The failure of proton pump inhibitors (PPIs) to completely resolve symptoms is an accepted problem, with approximately 25% of patients with GERD continuing to experience the symptoms of heartburn in spite of treatment. This study aims to demonstrate an earlier onset to relief of symptoms in patients suffering from heartburn associated with GERD using an immediate-release omeprazole/sodium bicarbonate formulation when compared with delayed-release omeprazole (Losec®).

ELIGIBILITY:
Inclusion Criteria:

Study patients will be included in the study if they satisfy the following criteria:

1. Male or female, between 18 and 75 years old.
2. History of frequent episodes of heartburn associated with GERD for at least 2 3 days per week during 2-4 weeks before screening and have responded to standard PPI therapy in the past 12 months.
3. Have not taken on-demand PPI therapy for > 3 consecutive days within 4 weeks before the screening period.
4. The patient's written informed consent must be obtained prior to inclusion.
5. Willing and able to complete the entire procedure and to comply with study instructions.
6. Females of childbearing potential must employ an adequate method of birth control.

Inclusion criteria applicable to Screening period:

1. Recorded at least 1 evaluable episode of heartburn on 2 separate days at level 4 or higher on the 9-point Likert severity scale (point 3 on a 0-8 point scale) prior to randomisation.
2. Competent in the use and completion of the e-diary.

Exclusion Criteria:

Study patients will be excluded if they meet any of the following criteria:

1. Age < 18 or > 75 years old.
2. Intake of any medication for the purpose of the eradication of Helicobacter pylori (H. pylori) during the last 28 days before the start of the study.
3. Intake of systemic glucocorticoids or non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2-inhibitors (≥ 3 consecutive days per week) during the last 28 days before the start of the study; except regular intake of enteric coated aspirin dosages up to 150 mg/d.
4. Previously underwent acid-lowering surgery or other surgery of the oesophagus and/or upper gastrointestinal tract (excluding: appendectomy, cholecystectomy and polypectomy).
5. History of co-existing disease that affects the oesophagus (e.g. Barrett's oesophagus, Zollinger-Ellison syndrome, oesophageal stricture), and have undergone an endoscopy with results of incomplete healing of erosions following standard PPI therapy within the last 3 months.
6. History of active gastric or duodenal ulcers within 3 months of the first dose of the study drug or had acute upper gastrointestinal (GI) bleeding within last 6 months.
7. Documented presence of severe renal or hepatic insufficiency.
8. Known hypersensitivity to omeprazole.
9. Concurrent participation in a study with an investigational drug or participation within 30 days of study entry.
10. Females who are pregnant, or planning a pregnancy. Females of child bearing potential not using reliable methods of birth control.
11. Clinically significant laboratory abnormality or disease which, in the opinion of the Investigator, will create a risk for the patient, obscure the effects of study treatment or interfere with study results.
12. Received or require any of the following drugs within 2 weeks before the first dose of study or continue to need these drugs for concurrent therapy: theophylline, bismuth salts, warfarin, phenytoin, tacrolimus, diazepam, cyclosporine, disulfiram, benzodiazepines, barbiturates, antineoplastic agents, erythromycin, clarithromycin, sucralfate, clopidogrel or protease inhibitors.
13. Taking concomitant medications that rely on the presence of gastric acid for optimal bioavailability (e.g. ketoconazole, ampicillin esters or iron salts).
14. Onset of psychoactive medication (e.g. depressants, stimulants or hallucinogens) in the previous 6 months and during the entire course of the study.

Exclusion criteria applicable to Screening period:

1. Recorded < 1 episode of heartburn on 2 separate days at level 4 on the 9 point Likert severity scale (point 3 on a 0-8 point scale) during the 7 day screening period prior to randomisation
2. Completing < 90% (< 9 out of 10) of the time points with evaluable data on the e diary.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Regula, MD, Principal Investigator — Dept of Gastroenterology and Hepatology, Roentgena, Warsaw, Poland
Locations (1):
- Department of Gastroenterology and Hepatology, Oncology Centre, Roentgena, Warsaw, Poland

REFERENCES:
- [Derived] Walker D, Ng Kwet Shing R, Jones D, Gruss HJ, Regula J. Challenges of correlating pH change with relief of clinical symptoms in gastro esophageal reflux disease: a phase III, randomized study of Zegerid versus Losec. PLoS One. 2015 Feb 23;10(2):e0116308. doi: 10.1371/journal.pone.0116308. eCollection 2015. PMID 25706883

RESULTS

PARTICIPANT FLOW:
Groups:
- Zegerid: Treatment of heartburn with 20mg Zegerid suspension plus over-encapsulated placebo capsule once a day
- Losec: Treatment of heartburn with 20mg Losec over-capsulated capsule plus placebo suspension once a day
Period: Overall Study
Arm/Group | Zegerid | Losec
Started | 122 | 117
Completed | 119 | 114
Not Completed | 3 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zegerid | Losec | Total
Number analyzed (Participants) | 122 | 117 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 110 | 219
  >=65 years | 13 | 7 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 45.0 (15.43) | 44.4 (13.91) | 44.7 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 69 | 131
  Male | 60 | 48 | 108
Region of Enrollment [Number; unit: participants]
  Poland | 48 | 49 | 97
  Bulgaria | 14 | 17 | 31
  Czech Republic | 17 | 15 | 32
  Hungary | 19 | 14 | 33
  Romania | 17 | 18 | 35
  United Kingdom | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Determination of Median Time to Sustained Partial Response as Defined by Reduction in Likert Severity Scale Used to Assess Pain Associated With Heartburn in the Patient
Description: Reduction in severity of heartburn by 2 points or more on a 9-point Likert severity scale, which is sustained for 45 minutes or more
Time Frame: up to 14 days following treatment
Population: mITT
Measure: Median (95% Confidence Interval); unit: Minutes
Groups:
- Zegerid Group: 20mg Zegerid suspension plus over-encapsulated placebo capsule
- Losec Group: 20mg Losec over-encapsulated capsule plus placebo suspension
Arm/Group | Zegerid Group | Losec Group
Number analyzed (Participants) | 117 | 111
Minutes | 37.5 [30.00 to 45.00] | 37.5 [30.00 to 45.00]
Statistical Analysis 1: Comparison: Zegerid Group vs Losec Group; Test type: Superiority or Other; p = 0.563, Regression, Cox; Hazard Ratio (HR) = 1.097

2. Secondary Outcome: Median Time to Sustained Partial Response
Description: as for outcome 1
Time Frame: up to 14 days
Population: mITT
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Zegerid Group | Losec Group
Number analyzed (Participants) | 117 | 111
Minutes | 37.5 [30.0 to 45.0] | 37.5 [30.0 to 45.0]
Statistical Analysis 1: Comparison: Zegerid Group vs Losec Group; Test type: Superiority or Other; p = 0.712, Regression, Cox; Hazard Ratio (HR) = 0.903

3. Secondary Outcome: Median Time to Sustained Total Relief
Description: Time to sustained total relief, defined as zero severity (no heartburn) on a 9-point Likert severity scale, which is sustained for 45 minutes or more
Time Frame: 14 days
Population: mITT
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Zegerid Group | Losec Group
Number analyzed (Participants) | 117 | 111
Minutes | 105.0 [90.0 to 120.0] | 105.0 [75.0 to 120.0]
Statistical Analysis 1: Comparison: Zegerid Group vs Losec Group; Test type: Superiority or Other; p = 0.457, Regression, Cox; Hazard Ratio (HR) = 1.140

4. Secondary Outcome: Percentage of Patients Responding in 45 Minutes
Description: percentage of patients who have achieved sustained partial response, sustained response, or sustained total relief, by 45 minutes
Time Frame: up to 14 days
Population: mITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Zegerid Group | Losec Group
Number analyzed (Participants) | 117 | 111
percentage of patients | 65 [55.6 to 73.5] | 62.2 [52.5 to 71.2]
Statistical Analysis 1: Comparison: Zegerid Group vs Losec Group; Sustained partial response; Test type: Superiority or Other; p = 0.625, Regression, Cox; Mean Difference (Final Values) = 2.8, 95% CI [-9.7 to 15.3]
Statistical Analysis 2: Comparison: Zegerid Group vs Losec Group; Sustained response; Test type: Superiority or Other; p = 0.755, Regression, Cox; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-15.0 to 10.6]
Statistical Analysis 3: Comparison: Zegerid Group vs Losec Group; Sustained total relief; Test type: Superiority or Other; p = 0.194, Regression, Cox; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-3.6 to 17.2]

5. Secondary Outcome: Percentage of Patients Responding in 60 Minutes
Description: Proportion of patients who have achieved sustained response, sustained partial response or sustained total relief by 60 minutes
Time Frame: 14 days
Population: mITT
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Zegerid Group | Losec Group
Number analyzed (Participants) | 117 | 111
Percentage of patients | 74.4 [65.5 to 82.0] | 78.4 [69.6 to 85.6]
Statistical Analysis 1: Comparison: Zegerid Group vs Losec Group; Sustained partial response; Test type: Superiority or Other; p = 0.501, Regression, Cox; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-15.0 to 7.0]
Statistical Analysis 2: Comparison: Zegerid Group vs Losec Group; Sustained response; Test type: Superiority or Other; p = 0.518, Regression, Cox; Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-17.6 to 8.2]
Statistical Analysis 3: Comparison: Zegerid Group vs Losec Group; Sustained total relief; Test type: Superiority or Other; p = 0.794, Regression, Cox; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-11.2 to 13.1]

6. Secondary Outcome: Percentage of Patients Responding in 90 Minutes
Description: Proportion of patients who have achieved sustained response, sustained partial response or sustained total relief by 90 minutes
Time Frame: 14 days
Population: mITT
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Zegerid Group | Losec Group
Number analyzed (Participants) | 117 | 111
Percentage of patients | 88.0 [80.7 to 93.3] | 85.6 [77.6 to 91.5]
Statistical Analysis 1: Comparison: Losec Group; Sustained partial response; Test type: Superiority or Other; p = 0.494, Regression, Cox; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-6.3 to 11.2]
Statistical Analysis 2: Comparison: Zegerid Group vs Losec Group; Sustained response; Test type: Superiority or Other; p = 0.751, Regression, Cox; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-14.7 to 9.1]
Statistical Analysis 3: Comparison: Zegerid Group vs Losec Group; Sustained total relief; Test type: Superiority or Other; p = 0.690, Regression, Cox; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-16.4 to 9.6]

ADVERSE EVENTS:
Arm/Group | Zegerid | Losec
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/117
Other Adverse Events (participants affected / at risk) | 4/122 | 4/117
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zegerid (N=122) | Losec (N=117)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
paronychia (Infections and infestations) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No